CLINICAL TRIAL: NCT02889692
Title: Study of Chinese Medicine Plus Targeted Therapy Maintenance Versus Targeted Therapy Maintenance in Advanced Pulmonary Adenocarcinoma: A Randomized Double-blind Controlled Clinical Trial
Brief Title: Clinical Study of Chinese Medicine Plus Targeted Therapy Maintenance in Advanced Pulmonary Adenocarcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Shanghai Chest Hospital (Other); Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Ling Xu, Principal Investigator, Shanghai University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LH127
Record Dates: First submitted 2016-07-25; First posted 2016-09-05 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2016-08

CONDITIONS: Cancer
Keywords: lung cancer; traditional Chinese medicine; maintenance therapy; targeted therapy
MeSH Terms: conditions — Neoplasms; Lung Neoplasms | interventions — Erlotinib Hydrochloride; Gefitinib; icotinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TCM granules plus EGFR-TKIs (Experimental): TCM granules: oral granules, "YiQiFang" or "YangYinFang" or "YiQiYangYinFang", four packages, twice a day, until progression or unacceptable toxicity; EGFR-TKIs: oral tablet, Gefitinib® 250mg daily or Erlotinib® 150mg daily or Icotinib® 125 mg three times a day，until progression or unacceptable toxicity.
  Interventions: Drug: YiQiFang; Drug: YangYinFang; Drug: YiQiYangYinFang; Drug: Erlotinib®; Drug: Gefitinib®; Drug: Icotinib®
- Placebo granules plus EGFR-TKIs (Placebo Comparator): Placebo granules: oral granules, which the taste and smell are similar to experimental TCM granules and has no therapeutic effect, four packages, twice a day, until progression or unacceptable toxicity; EGFR-TKIs: oral tablet, Gefitinib® 250mg daily or Erlotinib® 150mg daily or Icotinib® 125 mg three times a day until progression or unacceptable toxicity.
  Interventions: Drug: placebo granules; Drug: Erlotinib®; Drug: Gefitinib®; Drug: Icotinib®

INTERVENTIONS:
Drug: YiQiFang — Prescriptions formulated into TCM granules origin from Professor Liu Jia-xiang in Longhua hospital. Package of granules is made into three types with functions such as benefiting Qi, benefiting Yin and detoxication recipe.
  YiQiFang: Patients with Qi deficiency syndrome are administered two packages of each benefiting Qi and detoxication recipe, four packages, twice a day, until progression or unacceptable.
  Arms: TCM granules plus EGFR-TKIs
Drug: YangYinFang — Prescriptions formulated into TCM granules origin from Professor Liu Jia-xiang in Longhua hospital. Package of granules is made into three types with functions such as benefiting Qi, benefiting Yin and detoxication recipe.
  YangYinFang: Patients with Yin deficiency syndrome are administered two packages of each benefiting Yin and detoxication recipe, four packages, twice a day, until progression or unacceptable.
  Arms: TCM granules plus EGFR-TKIs
Drug: YiQiYangYinFang — Prescriptions formulated into TCM granules origin from Professor Liu Jia-xiang in Longhua hospital. Package of granules is made into three types with functions such as benefiting Qi, benefiting Yin and detoxication recipe.
  YiQiYangYinFang: Patients with Qi and Yin deficiency syndrome are administered one package of each benefiting Qi and benefiting Yin and two packages of detoxication recipe, four packages, twice a day, until progression or unacceptable.
  Arms: TCM granules plus EGFR-TKIs
Drug: placebo granules — Oral granules, which the taste and smell are similar to experimental TCM granules, has no therapeutic effect, four packages, twice a day, until progression or unacceptable.
  Arms: Placebo granules plus EGFR-TKIs
Drug: Erlotinib® — "Erlotinib®","tarceva", 150 mg oral once a day until progression or unacceptable toxicity develops.
  Other Names: tarceva
Drug: Gefitinib® — "Gefitinib®","Iressa", 250 mg oral once a day until progression or unacceptable toxicity develops.
  Other Names: Iressa
Drug: Icotinib® — "Icotinib®","Conmana" 125 mg oral three times a day until progression or unacceptable toxicity develops.
  Other Names: Conmana

SUMMARY:
The investigators performed a randomized, double blind controlled, prospective study method on observation of Traditional Chinese Medicine (TCM) combined with targeted therapy maintenance to prolong the efficacy of long-term survival of advanced pulmonary adenocarcinoma patients. The investigators plan to involve 200 cases for observation in 3 years (100 cases for targeted therapy maintenance, 100 cases for targeted therapy maintenance plus TCM,), expecting that integrated TCM combined with targeted maintenance therapy has a better efficacy on prolonging progression-free survival time, overall survival, improving quality of life(QOL) of patients than that of targeted maintenance therapy.

DETAILED DESCRIPTION:
Maintenance therapy refers to systemic therapy that may be given for patients with advanced NSCLC after 4 to 6 cycles of first-line chemotherapy. However, patients are only candidates for maintenance therapy if they have responded to their previous treatment or have stable disease and their tumors have not progressed. Epidermal growth factor receptor tyrosine kinase inhibitors (EGFRTKIs) such as Iressa and Erlotinib have proved effective in first or second line therapy for advanced pulmonary adenocarcinoma. Targeted therapy maintenance can be partly extend patient's TTP, but the toxicity and the side effects of targeted therapy will decrease QOL. Besides, high cost of targeted therapy will cause greater economic pressure on patients.The investigators' preliminary studies have shown that traditional Chinese medicine (TCM) can prolong survival time and improve QOL, but high-level evidences are needed.

The investigators perform a multicenter, randomized, double blind controlled, prospective study in advanced pulmonary adenocarcinoma patients with stage Ⅲ～Ⅳ. Advanced pulmonary adenocarcinoma patients after first-line chemotherapy will choose maintenance therapy according to the patient's wishes, including targeted therapy maintenance, chemotherapy maintenance and TCM maintenance therapy. Patients who choose targeted therapy maintenance are randomized over observational group (TCM granules plus targeted therapy maintenance),and control group (TCM placebo plus targeted therapy maintenance). The treatment should be continued until evidence of disease progression or unacceptable toxicity, and after that regular follow-up will be arranged. The primary efficacy assessments are: OS (overall survival); Secondary efficacy assessments are: (1) PFS (progression-free survival); (2) Objective response rate; (3) QOL (Functional Assessment of Cancer therapy-lung, FACT-L4.0 scales; Lung Cancer Symptom Scale, LCSS); (4) other efficacy assessments are: 1) TCM symptoms changes; 2) Toxicity, side effects and security of the treatments will be assessed at the same time. The investigators expect that integrated TCM combined with targeted therapy maintenance has a better efficacy on prolonging progression-free survival time, overall survival, improving QOL of patients than that of targeted therapy maintenance. Therefore the study can provide evidences for optimizing and promoting integrated TCM combined with Western Medicine treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically or cytologically confirmed of stage IIIa-IV pulmonary adenocarcinoma;
2. The efficacy evaluation of the first-line therapy is progression-free including complete response(CR), partial response(PR) and stable disease(SD);
3. Age ≥18 years old;
4. Physical status score (ECOG PS) ≤ 2 scores;
5. Estimated life expectancy of at least 12 weeks;
6. Participants have no major organ dysfunction: hemoglobin ≥9 g/dL, absolute neutrophil count (ANC) ≥1.5*109/L, platelets ≥100 *109/L,bilirubin ≤1.5ULN, alkaline phosphatase (AP), aspartate transaminase (AST) and alanine transaminase (ALT) ≤2.5 upper limited number(ULN) (AP, AST, ALT ≤5ULN is acceptable if liver has tumor involvement).INR≤1.5, APTT in the normal range( 1.2DLN-1.2ULN),creatinine ≤1.5ULN;
7. Planning for targeted maintenance.
8. Informed consent from the patient.

Exclusion Criteria:

1. The efficacy evaluation of the first-line therapy is progressive disease(PD);
2. Patient with other malignant tumor except NSCLC 5 years previous to study entry;
3. Patient has already received chemotherapy or other anticancer treatment;
4. Estimated life expectancy less than 12 weeks;
5. Brain metastasis (controlled brain metastasis and steroid free need is excluded);
6. History of cardiovascular disease: Congestive Heart Failure > grade II in NYHA.Unstable angina patients (have angina symptoms in rest) or a new occurrence of angina (began in the last 3 months) or myocardial infarction happens in the last 6 months;
7. Pregnant or child breast feeding women;
8. Mental or cognitive disorders;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-03; Primary Completion 2016-12-30 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | 2 months
  It referred to the interval time from the first date of randomization to that of death for any reason, the end of the study, or loss of follow-up.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 2 months
  Time from start of the study treatment to date of objective tumour progression (excluding clinical deterioration without evidence of objective progression).
Objective response rate (ORR) | 2 months
  The ORR (complete response (CR) plus partial response (PR)) was determined by the Response Evaluation Criteria In Solid Tumors (RECIST) (Eisenhauer et al, 2009) version 1.1.in Solid Tumors (RECIST1.1).
Quality of life (QOL) | 2 months
  QOL is assessed using Functional Assessment of Cancer therapy-lung (FACT-L) questionnaire .

OTHER OUTCOMES:
TCM symptoms changes | 2 months
  TCM symptoms changes are according to the lung cancer symptom classification quantization table in "Guiding Principles for Clinical Research of Traditional Chinese Medicine in the Treatment of Lung Cancer (2002 Edition)".
Safety assessment evaluated according to Common Toxicity Criteria | 2 months
  Safety assessment is evaluated according to Common Toxicity Criteria (CTC 3.0).

CONTACTS AND LOCATIONS:
Overall Officials: Ling c, MD & PhD, Principal Investigator — Longhua Hospital

IPD SHARING:
Plan to Share IPD: Yes